CLINICAL TRIAL: NCT03181581
Title: Improving Ultrasound Images in Brain Tumour Surgery With the Use of an Acoustic Coupling Fluid Mimicking Brain Tissue: a Phase II Technical and Safety Study
Brief Title: Improving Ultrasound Images in Brain Tumour Surgery With the Use of an Acoustic Coupling Fluid Mimicking Brain Tissue.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: because the study had to be redesigned and restarted as clinical device study
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian National Advisory Unit for Ultrasound and Image-guided Therapy (Unknown); SINTEF Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ACF-02; 2016-003025-42 (EudraCT Number)
Record Dates: First submitted 2017-06-02; First posted 2017-06-09 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Brain Neoplasms; Glioma
Keywords: ultrasonography; ultrasonics; brain; surgery
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Ringer's acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High grade gliomas stage 1 ACF (Experimental): In the first stage 12-15 patients with high-grade gliomas will be included in the trial (acoustic coupling fluid) group.
  Interventions: Biological: acoustic coupling fluid
- Low-high grade gliomas stage 2 ACF (Experimental): If the interim safety assessments validate that the study can continue, the second stage involves inclusion in the trial (acoustic coupling fluid) group of 22-25 patients with both low-grade and high-grade glioma
  Interventions: Biological: acoustic coupling fluid
- High grade gliomas stage 1 control (Active Comparator): In the first stage 12-15 patients with high-grade gliomas will be included in the Ringer's acetate (control) group.
  Interventions: Biological: Ringer's acetate
- Low-high grade gliomas stage 2 control (Active Comparator): If the interim safety assessments validate that the study can continue, the second stage involves inclusion in the Ringer's acetate (control) group of 22-25 patients with both low-grade and high-grade glioma
  Interventions: Biological: Ringer's acetate

INTERVENTIONS:
Biological: acoustic coupling fluid — ultrasound images obtained with both ACF and Ringer's acetate
  Other Names: ACF
  Arms: High grade gliomas stage 1 ACF; Low-high grade gliomas stage 2 ACF
Biological: Ringer's acetate — ultrasound images obtained with Ringer's acetate only
  Arms: High grade gliomas stage 1 control; Low-high grade gliomas stage 2 control

SUMMARY:
Tools for improving brain tumor surgery, in particular for gliomas, are increasing. There seems to be an agreement that achieving extensive resections, when done safely without jeopardizing neurological function, improves survival.

Ultrasound is currently used as a tool for providing 2D or 3D images for tumor localization and resection control. For the use in resection control the resection cavity is filled with saline to provide acoustic coupling between the ultrasound transducer and tissue. However, attenuation of acoustic waves is very low in saline compared to the brain and this difference in attenuation is the cause of artifacts that may severely degrade the ultrasound images. Such artifacts are seen as high-intensity signal at the resection cavity wall and beyond. The artificial signal enhancement can potentially mask small tumor remnants and is generally making the interpretation of images more difficult.

This research group has developed an acoustic coupling fluid intended for use in the resection cavity instead of saline. Tests in laboratory measurements have shown that the fluid reduces artifacts and has the potential to enhance ultrasound image quality in brain tumor surgery. Three different concentrations of the acoustic coupling fluid have been tested in a phase 1 study that included 15 patients with glioblastoma. The concentration that provided the optimal ultrasound images, from qualitative and quantitative inspection, is used in the current phase II study. This study is a randomized controlled trial aiming to include 82 patients with glial brain tumours. Its purpose is to test the fluid during surgery of glial brain tumours to further investigate safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* A diffuse glial tumour (high-grade (stage 1), low-grade or high-grade (stage 2)) is suspected from the diagnostic magnetic resonance images (MRI).
* In cases where histopathology is not known from previous biopsy or resection (i.e. diagnosis is suspected based on MRI findings and not from previous surgery) a tissue sample for frozen section is necessary to confirm the diagnosis.
* Karnofsky performance status >=70

Exclusion Criteria:

* Not able to consent (e.g. severe cognitive impairment)
* Intended biopsy only (meaning: cases not suitable for resection)
* Hypersensitivity to egg protein
* Hypersensitivity to soya or peanut protein
* Hypersensitivity to glycerol
* Pregnancy of breast-feeding
* Intention to become pregnant during the time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
difference in serious adverse event rates (test minus control) | 72 hours
  Non-inferiority (i.e. test serious adverse event rate is "not worse" than control) is shown if the 95%-confidence interval around the mean difference in event rates has an upper value below 0.3 which is the predefined margin
difference in serious adverse event rates (test minus control) | 30 days
  Non-inferiority (i.e. test serious adverse event rate is "not worse" than control) is shown if the 95%-confidence interval around the mean difference in event rates has an upper value below 0.3 which is the predefined margin
difference in serious adverse event rates (test minus control) | 6 months
  Non-inferiority (i.e. test serious adverse event rate is "not worse" than control) is shown if the 95%-confidence interval around the mean difference in event rates has an upper value below 0.3 which is the predefined margin

SECONDARY OUTCOMES:
image artefacts | 1 day
  during the operation; Qualitative score of ultrasound image quality (poor-medium-good)
image artefacts | 1 day
  during the operation; Qualitative score of artefacts in ultrasound images (none-some-much)
depiction of outline of the anatomy surrounding the resection cavity | 1 day
  during the operation; Qualitative score of ultrasound image quality (poor-medium-good)
depiction of outline of the anatomy surrounding the resection cavity | 1 day
  during the operation; Qualitative score of artefacts in ultrasound images (none-some-much)
image signal-to-noise ratio | 1 day
  after the operation: image analysis by quantitative measurements of signal-to-noise ratio (SNR)

OTHER OUTCOMES:
Quality of Life | 1 month
  assessed by EQ5D (generic)
Quality of Life | 1 month
  assessed by QLQ-C30 (cancer specific)
Quality of Life | 6 months
  assessed by EQ5D (generic)
Quality of Life | 6 months
  assessed by QLQ-C30 (cancer specific)

CONTACTS AND LOCATIONS:
Overall Officials: Petter Aadahl, phd md, Study Director — St. Olavs Hospital
Locations (1):
- Department of Neurosurgery, St Olavs Hospital, Trondheim, Norway